CLINICAL TRIAL: NCT03315351
Title: Feasibility of PET-scan Carried Out at Day 1 of Brachytherapy for Patients With Locally Advanced Cervical Cancer Treated Initially by Concomitant Radio-chemotherapy
Brief Title: Feasibility of Pet-scan at Day 1 of Brachytherapy for Patients With Cervical Cancer
Acronym: TEP-Curie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TEP-Curie-1702; 2017-A01888-45 (Other: ANSM)
Record Dates: First submitted 2017-09-25; First posted 2017-10-20 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Cervical Cancer
Keywords: PET-scan; Brachytherapy; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Procedure (Experimental): Brachytherapy. PET-scan.
  Interventions: Procedure: Brachytherapy; Other: PET-scan

INTERVENTIONS:
Procedure: Brachytherapy — Before it starts, a consultation will be done to collect patient's informations and disease history, a clinical exam will be done and an evaluation of radio-chemotherapy toxicity will be realized.
  The brachytherapy include a pulsating flow treatment driven by RMI and CT-scan
Other: PET-scan — The patient will undergo 2 PET-scan during the clinical trial:
  * the first one is additional to the brachytherapy
  * the second one is realized 4 months after the brachytherapy

SUMMARY:
Interventional, exploratory, prospective and monocentric study which aim to study the feasibility of brachytherapy using a PET-scan

DETAILED DESCRIPTION:
The study will proceed as follow:

* Initial check-up before the brachytherapy, including a clinical exam, collect of disease history and other informations that can be required for a good execution of the trial, and a usual patient care (chemotherapy with concomitant radiotherapy, biopsy, RMI, PET-scan and paraaortic lymphadenectomy).
* additional PET-scan exam at day 1 of the brachytherapy (with collect of informations on toxicity, clinical morphology data and biomorphological data of RMI and PET-scan, and dosimetric study of the brachytherapy)
* 4 months after the brachytherapy, additional PET-scan monitoring metabolic volumes and standardized metabolic fixation parameters

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from a cervical cancer:
* squamous-cell carcinoma or adenocarcinoma histologically proven
* classified from FIGO 2009 IB2 to IVA stage
* Age ≥ 18 years old
* Examination by PET-scan and pelvic RMI realized at diagnosis
* Examination by negative PET-scan remotely closed and at lymph node level
* Surgical lymphadenectomy negative at paraaortic level
* Treatment by external radiotherapy (doses between 45 Gy and 50.4 Gy in 1.8 Gy/fractions) and concomitant chemotherapy (at least 4 cures per weeks using platinum salt) done
* Scheduled curative treatment by brachytherapy driven by RMI
* Affiliation to the National Social Security System
* With informed and signed consent before any procedure specific to the study

Exclusion Criteria:

* Performance status of WHO score > 2
* Other histology than squamous cell carcinoma or adenocarcinoma
* Metastatic patient or paraaortic node positive
* Adjuvant radiochemotherapy after the first surgery
* Dementia or psychiatric history
* Kidney failure
* Diabet
* Chronic inflammatory bowel disease
* Pelvic and/or vesicoureteral surgery history
* Pelvic irradiation history
* Other active neoplasia or < 5 years old, except for basocellular carcinoma that can be locally treated
* Contraindication to one of the following procedure : RMI, PET-scan, general anesthesia
* Radiosensitive disease (Fragile X syndrome, Huntington's chorea, Xeroderma Pigmentosum, connective tissue disease) or signs of radiosensitivity.
* Treatment with palliative intent
* Pregnant or breastfeeding women
* Patient Under guardianship or tutorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of "TEP-Curie" (Brachytherapy driven by PET-scan) in terms of realized exams | 4 months
  Concerning this outcome, the success in terms of feasibility will be the possibility of realizing the TEP-Curie exam
Feasibility of "TEP-Curie" (Brachytherapy driven by PET-scan) regarding the possibility to define HR-CTV target volume (High-Risk Clinical Target Volume) | 4 months
  Concerning this outcome, the success in terms of feasibility will be the possibility of defining a HR-CTV target volume for at least one of the 3 proposed approaches using the PET
Feasibility of "TEP-Curie" (Brachytherapy driven by PET-scan) regarding the dicom medical image transfer | 4 months
  Concerning this outcome, the success in terms of feasibility will be the possibility of transfering image in a Dicom format
Feasibility of "TEP-Curie" (Brachytherapy driven by PET-scan) regarding the contouring possibility | 4 months
  Using the possibility of defining the contouring for at least one of the 3 alternative treatment plans

SECONDARY OUTCOMES:
Impact of the "TEP-Curie" (Brachytherapy driven by PET-scan) on target volume definition | 4 months
  Comparison of the target volume obtained with TEP-curie to the target volume defined by the RMI alone
Assessment of the HR-CTV coverage | 4 months
  Comparison of the HR-CTV obtained with TEP-curie to the HR-CTV obtained by the RMI alone
Assessment of the dose received by the neighboring target organs | 4 months
  Comparison of the dose obtained with TEP-curie to the dose obtained by the RMI alone
Time needed to design the different alternative treatment plans | 4 months
Toxicity linked to the standard treatment driven by RMI only | 4 months
  Graded according to the NCI CTCAE v4. scale

CONTACTS AND LOCATIONS:
Overall Officials: Abel CORDOBA, MD, Principal Investigator — Centre oscar Lambret de Lille
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No